CLINICAL TRIAL: NCT02236000
Title: A Phase Ib/II Dose-Escalation Study Evaluating the Combination of Trastuzumab Emtansine (T-DM1) With Neratinib in Women With Metastatic HER2-Positive Breast Cancer
Brief Title: A Dose-Escalation Study Evaluating the Combination of Trastuzumab Emtansine (T-DM1) With Neratinib in Women With Metastatic HER2-Positive Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NSABP Foundation Inc (Network)
Collaborators: Puma Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSABP FB-10
Record Dates: First submitted 2014-09-02; First posted 2014-09-10 (Estimated); Results first posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Breast Cancer
Keywords: NSABP; Trastuzumab Emtansine; T DM1; Neratinib; Metastatic Breast Cancer; HER2 positive; Dose Escalation
MeSH Terms: conditions — Breast Neoplasms | interventions — neratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Neratinib and T-DM1 (Experimental)
  Interventions: Drug: Neratinib; Drug: T-DM1

INTERVENTIONS:
Drug: Neratinib — Dose-Escalation Phase (Part 1) - Neratinib Dose-escalation will proceed on the basis of DLT during Cycle 1 starting at 120 mg/day.
  Dose level 1: 120 mg/day; Dose level 2: 160 mg/day; Dose level 3: 200 mg/day; Dose level 4: 240 mg/day
  Dose-evaluation Phase (Part 2) - Patients will receive the highest dose of neratinib with T-DM1 found in Phase I as study therapy
Drug: T-DM1 — Dose-Escalation Phase (Part 1) - Trastuzumab emtansine (T-DM1) will be given at 3.6 mg/kg IV Day 1 every 21 days.
  Dose-evaluation Phase (Part 2) - Trastuzumab emtansine (T-DM1) will be given at 3.6 mg/kg IV Day 1 every 21 days.

SUMMARY:
This study is being done for the following reasons:

* The study has two parts. The purpose of the first part (Phase I) of the study is to find out the highest dose of neratinib that can be given safely with T-DM1.
* The purpose of the second part of the study (Phase II) is to find out whether the dose of neratinib with T-DM1 determined in Phase I will keep breast cancer from getting worse for a period of time.
* In order to learn more about study therapy levels in blood and discover genetic and protein changes associated with cancer, the study includes special research tests using samples from blood and from breast tumor. Blood samples will be collected before study treatment, once during treatment, and after study treatment stops.
* In the optional part of this study, three biopsies will be performed to obtain fresh tumor samples from an area where your cancer has spread.

DETAILED DESCRIPTION:
The FB-10 study is designed as an open label, single arm, Phase Ib/II study with a dose-escalation phase and an expanded cohort (phase II) to evaluate the combination of trastuzumab emtansine (T-DM1) with neratinib in women with metastatic, HER2-positive breast cancer. The primary aim of the phase Ib portion of this study is to determine the safety and tolerability of the two-drug combination. The primary aim of the phase II portion is to demonstrate efficacy.

Patients will receive concurrent therapy with T-DM1 (3.6 mg/kg IV) on Day 1 of a 3-week (21 day) cycle and neratinib as a continuous daily oral dose. The neratinib dose-escalation will include 4 dose levels (120 mg, 160 mg, 200 mg, and 240 mg). At the recommended phase II dose (RP2D) of the T-DM1 and neratinib combination, up to 39 additional patients will be treated.

The sample size of the phase I portion of the study was 27 patients. The sample size of the Phase II portion will be 22 evaluable patients (and 4 replacement patients). The total study enrollment, phase Ib and II, will be a maximum of 50 patients.

Submission of diagnostic tumor samples and blood samples for FB-10 correlative science studies will be a study requirement for all patients. Blood samples for pharmacokinetics (PKs) and for future study will be collected prior to administration of study therapy on Cycle 1/Day 1, Cycle 1/Day 8, and Cycle 2/Day1.

A tumor biopsy will be procured from an accessible site of metastasis before study therapy is initiated (after the patient has signed the consent and has been screened for eligibility).

ELIGIBILITY:
Inclusion Criteria:

* The ECOG performance status must be less than or equal to 2.
* Patients must have the ability to swallow oral medication.
* Patients must have histologic or cytologic confirmation of the diagnosis of invasive adenocarcinoma of the breast.
* Patients must have had anti-HER2 based therapy with pertuzumab and trastuzumab for neoadjuvant therapy, adjuvant therapy or with first line therapy for metastatic disease (which may include trastuzumab and pertuzumab either sequentially or in combination).
* There must be documentation that the patient has evidence of measurable metastatic breast cancer that is accessible to biopsy at study entry.
* Patients must have estrogen receptor (ER) analysis performed prior to study entry. If ER analysis is negative, then progesterone receptor (PgR) analysis must also be performed. (Patients are eligible with either hormone receptor-positive or hormone receptor-negative tumors.)
* Breast cancer must be determined by local testing to be human epidermal growth factor receptor 2 (HER2)-positive prior to study entry using American Society of Clinical Oncology (ASCO) - College of American Pathologists (CAP) HER2 test guidelines.
* At the time of study entry, blood counts performed within 4 weeks prior to study entry must meet the following criteria:

  * absolute neutrophil count (ANC) must be greater than or equal to 1000/mm3;
  * platelet count must be greater than or equal to 100,000/mm3; and
  * hemoglobin must be greater than or equal to 9 g/dL. (Note: Patient must have discontinued growth factors greater than or equal to two weeks prior to entry labs.)
* The following criteria for evidence of adequate hepatic function performed within 4 weeks prior to study entry must be met:

  * Total bilirubin must be less than or equal to 1.5 x upper limit of normal (ULN), and
  * aspartate aminotransferase (AST) and alanine aminotransferase (ALT) must be less than or equal to 1.5 x ULN for the lab or less than or equal to 5 x ULN if liver metastasis.
* Serum creatinine performed within 4 weeks prior to study entry must be less than or equal to 1.5 x ULN for the lab.
* The left ventricular ejection fraction (LVEF) assessment by 2-D echocardiogram or multi-gated acquisition (MUGA) scan performed within 90 days prior to study entry must be greater than or equal to 50% regardless of the facility's lower limit of normal (LLN).
* Patients with reproductive potential must agree to use an effective non-hormonal method of contraception during therapy, and for at least 7 months after the last dose of study therapy.

Exclusion Criteria

* Previous therapy with T-DM1 or any HER2 tyrosine kinase inhibitor (TKI) including neratinib for any malignancy.
* Symptomatic brain metastases or brain metastases requiring chronic steroids to control symptoms.
* Active hepatitis B or hepatitis C with abnormal liver function tests; HIV positive patients receiving antivirals.
* Lung disease resulting in dyspnea at rest.
* Active infection or chronic infection requiring chronic suppressive antibiotics.
* Malabsorption syndrome, ulcerative colitis, inflammatory bowel disease, resection of the stomach or small bowel, or other disease or condition significantly affecting gastrointestinal function.
* Persistent greater than or equal to grade 2 diarrhea regardless of etiology.
* Conditions that would prohibit intermittent administration of corticosteroids for T-DM1 premedication.
* Chronic daily treatment with corticosteroids with a dose of greater than or equal to 10 mg/day methylprednisolone equivalent (excluding inhaled steroids).
* Uncontrolled hypertension defined as a systolic BP greater than 150 mmHg or diastolic BP greater than 90 mmHg, with or without anti-hypertensive medications. (Patients with hypertension that is well controlled on medication are eligible.)
* Cardiac disease (history of and/or active disease) that would preclude the use of any of the drugs included in the treatment regimen. This includes but is not confined to:

  * Active cardiac disease: symptomatic angina pectoris within the past 90 days that required the initiation of or increase in anti-anginal medication or other intervention; ventricular arrhythmias except for benign premature ventricular contractions; supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medication; conduction abnormality requiring a pacemaker; valvular disease with documented compromise in cardiac function; and symptomatic pericarditis
  * History of cardiac disease: myocardial infarction documented by elevated cardiac enzymes or persistent regional wall abnormalities on assessment of left ventricular (LV) function; history of documented congestive heart failure (CHF); and documented cardiomyopathy
* Other nonmalignant systemic disease that would preclude the patient from receiving study treatment or would prevent required follow up.
* Pregnancy or lactation at the time of study entry. (Note: Pregnancy testing should be performed within 14 days prior to study entry according to institutional standards for women of childbearing potential.)
* The investigator should assess the patient to determine if she has any psychiatric or addictive disorder or other condition that, in the opinion of the investigator, would preclude her from meeting the study requirements.
* Use of any investigational agent within 4 weeks prior to study entry.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2014-08; Primary Completion 2020-12 (Actual); Study Completion 2021-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — NSABP Foundation Inc
Locations (15):
- United States (15):
  - Cleveland Clinic Weston, Weston, Florida
  - Cancer Care Specialists of Central Illinois, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Cancer Care Specialists of Central Illinois-Swansea, Swansea, Illinois
  - Cleveland Clinic, Cleveland, Ohio
  - Stephenson Cancer Center at the University of Oklahoma Health Services Center, Oklahoma City, Oklahoma
  - UPMC- Hillman Cancer Center-Monroeville, Monroeville, Pennsylvania
  - Alleheny General Hospital, Pittsburgh, Pennsylvania
  - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Magee Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - UPMC- St. Margaret, Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center North Hills at Passavant, Pittsburgh, Pennsylvania
  - Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - West Virginia University, Morgantown, West Virginia

REFERENCES:
- [Derived] Jacobs SA, Wang Y, Abraham J, Feng H, Montero AJ, Lipchik C, Finnigan M, Jankowitz RC, Salkeni MA, Maley SK, Puhalla SL, Piette F, Quinn K, Chang K, Nagy RJ, Allegra CJ, Vehec K, Wolmark N, Lucas PC, Srinivasan A, Pogue-Geile KL. NSABP FB-10: a phase Ib/II trial evaluating ado-trastuzumab emtansine (T-DM1) with neratinib in women with metastatic HER2-positive breast cancer. Breast Cancer Res. 2024 Apr 22;26(1):69. doi: 10.1186/s13058-024-01823-8. PMID 38650031
- [Derived] Abraham J, Montero AJ, Jankowitz RC, Salkeni MA, Beumer JH, Kiesel BF, Piette F, Adamson LM, Nagy RJ, Lanman RB, Sperinde J, Huang W, Allegra CJ, Srinivasan A, Wang Y, Pogue-Geile KL, Lucas PC, Jacobs SA. Safety and Efficacy of T-DM1 Plus Neratinib in Patients With Metastatic HER2-Positive Breast Cancer: NSABP Foundation Trial FB-10. J Clin Oncol. 2019 Oct 10;37(29):2601-2609. doi: 10.1200/JCO.19.00858. Epub 2019 Aug 23. PMID 31442103

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase 1 consisted of 4 parts involving increasing doses of Neratinib in each part. Together, 27 patients were enrolled. In Phase II, 22 patients were enrolled. Therefore 49 patients were enrolled in both phases of the trial.
Pre-assignment Details: Endpoint information is not available for 1 patient.
Groups:
- Phase 1-Neratinib 120mg; T-DM1 3.6mg/kg: Dose Level 1- Neratinib 120mg T-DM1 3.6.mg/kg
- Phase 1-Neratinib 160 mg; T-DM1 3.6mg/kg: Dose Level 2- Neratinib 160 mg T-DM1 3.6mg/kg
- Phase 1-Neratinib 200mg; T-DM1 3.6mg/kg: Dose Level 3- Neratinib 200mg T-DM1 3.6mg/kg
- Phase 1 Neratinib 240; T-DM1 3.6mg/kg: Dose Level 4- Neratinib 240mg T-DM1 3.6 mg/kg
- Neratinib and T-DM1 Part 2 (Phase II): Dose-evaluation Phase (Part 2)-Patients will receive the highest dose of neratinib with T-DM1 found in Phase I as study therapy. Dose-evaluation Phase (Part 2)-Trastuzumab ematansine (T-DM1) will be given at 3.6 mg/kg IV Day 1 ever 21 days.
Period: Overall Study
Arm/Group | Phase 1-Neratinib 120mg; T-DM1 3.6mg/kg | Phase 1-Neratinib 160 mg; T-DM1 3.6mg/kg | Phase 1-Neratinib 200mg; T-DM1 3.6mg/kg | Phase 1 Neratinib 240; T-DM1 3.6mg/kg | Neratinib and T-DM1 Part 2 (Phase II)
Started | 6 | 10 | 8 | 3 | 22
Completed | 6 | 10 | 8 | 3 | 22
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase 1-Neratinib 120mg; T-DM1 3.6mg/kg: Dose Level 1-Neratinib 120mg T-DM1 3.6mg/kg
- Phase 1-Neratinib160mg; T-DM1 3.6mg/kg: Dose Level 2-Neratinib 160mg T-DM1 3.6mg/kg
- Phase 1-Neratinib 200mg; T-DM1 3.6mg/kg: Dose Level 3-Neratinib 200mg T-DM1 3.6 mg/kg
- Phase 1 Neratinib 240mg; T-DM1 3.6mg/kg: Dose Level 4-Neratinib 240mg T-DM1 3.6mg/kg
- Neratinib and T-DM1 Part 2 (Phase II): Dose-evaluation Phase (Part 2) - Patients will receive the highest dose of neratinib with T-DM1 found in Phase I as study therapy.
  Dose-evaluation Phase (Part 2) - Trastuzumab emtansine (T-DM1) will be given at 3.6 mg/kg IV Day 1 every 21 days.
- Total: Total of all reporting groups
Arm/Group | Phase 1-Neratinib 120mg; T-DM1 3.6mg/kg | Phase 1-Neratinib160mg; T-DM1 3.6mg/kg | Phase 1-Neratinib 200mg; T-DM1 3.6mg/kg | Phase 1 Neratinib 240mg; T-DM1 3.6mg/kg | Neratinib and T-DM1 Part 2 (Phase II) | Total
Number analyzed (Participants) | 6 | 10 | 8 | 3 | 22 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (15.30) | 51.1 (13.24) | 51.0 (9.40) | 42.0 (7.00) | 55.5 (10.35) | 52.08 (11.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 8 | 3 | 22 | 49
  Male | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 2 | 3
  Not Hispanic or Latino | 6 | 9 | 8 | 3 | 20 | 46
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 1 | 0 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 0 | 0 | 2
  White | 6 | 6 | 6 | 3 | 20 | 41
  More than one race | 0 | 2 | 1 | 0 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Evaluable Patients With Dose Limiting Toxicity Events in Phase 1
Description: If 1 of 3 patients in this cohort experiences a dose limiting toxicity (DLT), 3 more patients will be added at the same dose level. If 0 of 3 initial patients or 1 of 6 patients in an expanded cohort experiences a DLT, the dose for the next cohort will be escalated to dose level 2; otherwise, the combination will be considered too toxic.
Time Frame: Day 1, 8, and 15 of cycle 1.
Population: ITT patients who are evaluable for toxicity during the 1st cycle (patients who completed Cycle 1 or had a DLT) of the Phase 1 portion of the study.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1 Neratinib 120mg; T-DM1 3.6mg/kg: Dose Level 1-Neratinib 120mg T-DM1 3.6mg/kg
- Phase 1 Neratinib 160mg; T-DM1 3.6mg/kg: Dose Level 2-Neratinib 160mg T-DM1 3.6mg/kg
- Phase 1 Neratinib 200mg; T-DM1 3.6mg/kg: Dose Level 3-Neratinib 200mg T-DM1 3.6mg/kg
- Neratinib and T-DM1: Neratinib: Dose-Escalation Phase (Part 1) - Neratinib Dose-escalation will proceed on the basis of DLT during Cycle 1 starting at 120 mg/day.
  Dose level 1: 120 mg/day; Dose level 2: 160 mg/day; Dose level 3: 200 mg/day; Dose level 4: 240 mg/day
  Dose-evaluation Phase (Part 2) - Patients will receive the highest dose of neratinib with T-DM1 found in Phase I as study therapy
  T-DM1: Dose-Escalation Phase (Part 1) - Trastuzumab emtansine (T-DM1) will be given at 3.6 mg/kg IV Day 1 every 21 days.
  Dose-evaluation Phase (Part 2) - Trastuzumab emtansine (T-DM1) will be given at 3.6 mg/kg IV Day 1 every 21 days.
Arm/Group | Phase 1 Neratinib 120mg; T-DM1 3.6mg/kg | Phase 1 Neratinib 160mg; T-DM1 3.6mg/kg | Phase 1 Neratinib 200mg; T-DM1 3.6mg/kg | Phase 1 Neratinib 240mg; T-DM1 3.6mg/kg | Neratinib and T-DM1
Number analyzed (Participants) | 6 | 9 | 8 | 3 | 26
Participants | 1 | 0 | 4 | 2 | 7

2. Primary Outcome: Overall Response Rate (ORR) by Measurement of Target Lesions in Phase II
Description: Per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Every 42 days after the start of protocol therapy through disease progression, approximately 2 years
Population: ITT poplulation
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Neratinib and T-DM1: Dose-evaluation Phase (Part 2) - Patients will receive the highest dose of neratinib with T-DM1 found in Phase I as study therapy
  Dose-evaluation Phase (Part 2) - Trastuzumab emtansine (T-DM1) will be given at 3.6 mg/kg IV Day 1 every 21 days.
Arm/Group | Neratinib and T-DM1
Number analyzed (Participants) | 22
percentage of participants | 31.8 [15.99 to 51.55]

3. Secondary Outcome: Progression-free Survival (PFS) Time From Start of Study Therapy to Disease Progression or Death From Any Cause
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Every 42 days after the start of protocol therapy through disease progression, approximately 2 years
Population: ITT population
Measure: Median (95% Confidence Interval); unit: weeks
Groups:
- Neratinib and T-DM1 Part 1 (Phase I): Neratinib: Dose-Escalation Phase (Part 1) - Neratinib Dose-escalation will proceed on the basis of DLT during Cycle 1 starting at 120 mg/day.
  Dose level 1: 120 mg/day; Dose level 2: 160 mg/day; Dose level 3: 200 mg/day; Dose level 4: 240 mg/day
  T-DM1: Dose-Escalation Phase (Part 1) - Trastuzumab emtansine (T-DM1) will be given at 3.6 mg/kg IV Day 1 every 21 days.
Arm/Group | Phase 1 Neratinib 120mg; T-DM1 3.6mg/kg | Phase 1 Neratinib 160mg; T-DM1 3.6mg/kg | Phase 1 Neratinib 200mg; T-DM1 3.6mg/kg | Phase 1 Neratinib 240mg; T-DM1 3.6mg/kg | Neratinib and T-DM1 Part 1 (Phase I) | Neratinib and T-DM1 Part 2 (Phase II)
Number analyzed (Participants) | 6 | 10 | 8 | 3 | 27 | 22
weeks | 40 [22.00 to 72.29] | 15.4 [2.00 to NA] — Small sample size results in infinite upper 95% confidence bound. | 8.86 [3.00 to 80.00] | 9.00 [0.00 to NA] — Small sample size results in infinite upper 95% confidence bound. | 22 [3.29 to NA] — Small sample size results in infinite upper 95% confidence bound. | 27 [8 to 61]

4. Secondary Outcome: Adverse Events Experienced by Participants as a Measure of Toxicity
Description: Summary of frequency and severity of serious adverse events,
Time Frame: Day 1, 8, 15 of cycle one, day 1 of each subsequent cycle, at the end of protocol therapy and 30 days following the end of protocol therapy. Duration of therapy varied across patients from a few days to a couple of years.
Population: ITT population
Measure: Count of Participants; unit: Participants
Groups:
- Neratinib and T-DM-1 Part 2 (Phase 2): Dose-evaluation Phase (Part 2) - Patients will receive the highest dose of neratinib with T-DM1 found in Phase I as study therapy.
  Dose-evaluation Phase (Part 2) - Trastuzumab emtansine (T-DM1) will be given at 3.6 mg/kg IV Day 1 every 21 days.
Arm/Group | Phase 1 Neratinib 120mg; T-DM1 3.6mg/kg | Phase 1 Neratinib 160mg; T-DM1 3.6mg/kg | Phase 1 Neratinib 200mg; T-DM1 3.6mg/kg | Phase 1 Neratinib 240mg; T-DM1 3.6mg/kg | Neratinib and T-DM-1 Part 2 (Phase 2)
Number analyzed (Participants) | 6 | 10 | 8 | 3 | 22
Participants | 1 | 3 | 3 | 0 | 10

5. Secondary Outcome: Clinical Benefit Rate (Phase II)
Description: Per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.0) for target lesions assessed by MRI or CT; Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of new lesions; Stable Disease (SD) otherwise; Clinical Benefit (CB) = CR+PR+SD (confirmation of response not required).
Time Frame: Every 63 days after the start of study therapy until disease progression or until 30 days following the end of protocol therapy if due to another cause. Duration of therapy varied across patients from a few days to a couple of years.
Population: ITT population
Measure: Count of Participants; unit: Participants
Groups:
- Neratinib and T-DM1: Dose-evaluation Phase (Part 2) - Patients will receive the highest dose of neratinib with T-DM1 found in Phase I as study therapy.
  Dose-evaluation Phase (Part 2) - Trastuzumab emtansine (T-DM1) will be given at 3.6 mg/kg IV Day 1 every 21 days.
Arm/Group | Neratinib and T-DM1
Number analyzed (Participants) | 22
Participants | 12

ADVERSE EVENTS:
Time Frame: From cycle 1 day 1 until 30 days after the end of protocol therapy (or start of new therapy if it occurred before). The duration of therapy varied across patients from a few days to a couple of years as it was to be given until disease progression or intolerable toxicity.
Groups:
- Phase 1 Neratinib 120mg; T-DM1 3.6mg/kg: Neratinib 120mg T-DM1 3.6mg/kg
- Phase 1 Neratinib 160mg; T-DM1 3.6mg/kg: Neratinib 160mg T-DM1 3.6mg/kg
- Phase 1 Neratinib 200mg; T-DM1 3.6mg/kg: Neratinib 200mg T-DM1 3.6mg/kg
- Phase 1 Neratinib 240mg; T-DM1 3.6mg/kg: Neratinib 240mg T-DM1 3.6mg/kg
- Neratinib and T-DM1 Part 1 (Phase 1): Neratinib: Dose-Escalation Phase (Part 1) - Neratinib Dose-escalation will proceed on the basis of DLT during Cycle 1 starting at 120 mg/day.
  Dose level 1: 120 mg/day; Dose level 2: 160 mg/day; Dose level 3: 200 mg/day; Dose level 4: 240 mg/day
  T-DM1: Dose-Escalation Phase (Part 1) - Trastuzumab emtansine (T-DM1) will be given at 3.6 mg/kg IV Day 1 every 21 days.
- Neratinib and T-DM1Part 1 (Phase 2): Dose-evaluation Phase (Part 2) - Patients will receive the highest dose of neratinib with T-DM1 found in Phase I as study therapy.
  Dose-evaluation Phase (Part 2) - Trastuzumab emtansine (T-DM1) will be given at 3.6 mg/kg IV Day 1 every 21 days.
Arm/Group | Phase 1 Neratinib 120mg; T-DM1 3.6mg/kg | Phase 1 Neratinib 160mg; T-DM1 3.6mg/kg | Phase 1 Neratinib 200mg; T-DM1 3.6mg/kg | Phase 1 Neratinib 240mg; T-DM1 3.6mg/kg | Neratinib and T-DM1 Part 1 (Phase 1) | Neratinib and T-DM1Part 1 (Phase 2)
All-Cause Mortality (participants affected / at risk) | 0/6 | 1/10 | 0/8 | 0/3 | 1/27 | 1/22
Serious Adverse Events (participants affected / at risk) | 1/6 | 3/10 | 3/8 | 0/3 | 7/27 | 10/22
Other Adverse Events (participants affected / at risk) | 6/6 | 10/10 | 8/8 | 3/3 | 27/27 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Neratinib 120mg; T-DM1 3.6mg/kg (N=6) | Phase 1 Neratinib 160mg; T-DM1 3.6mg/kg (N=10) | Phase 1 Neratinib 200mg; T-DM1 3.6mg/kg (N=8) | Phase 1 Neratinib 240mg; T-DM1 3.6mg/kg (N=3) | Neratinib and T-DM1 Part 1 (Phase 1) (N=27) | Neratinib and T-DM1Part 1 (Phase 2) (N=22)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthritis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Neratinib 120mg; T-DM1 3.6mg/kg (N=6) | Phase 1 Neratinib 160mg; T-DM1 3.6mg/kg (N=10) | Phase 1 Neratinib 200mg; T-DM1 3.6mg/kg (N=8) | Phase 1 Neratinib 240mg; T-DM1 3.6mg/kg (N=3) | Neratinib and T-DM1 Part 1 (Phase 1) (N=27) | Neratinib and T-DM1Part 1 (Phase 2) (N=22)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 9 (9) | 7 (7) | 3 (3) | 25 (25) | 19 (19)
Nausea (Gastrointestinal disorders) | 6 (6) | 6 (6) | 3 (3) | 3 (3) | 18 (18) | 9 (9)
Constipation (Gastrointestinal disorders) | 4 (4) | 4 (4) | 4 (4) | 0 (0) | 12 (12) | 8 (8)
Vomiting (Gastrointestinal disorders) | 3 (3) | 5 (5) | 4 (4) | 1 (1) | 13 (13) | 7 (7)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 5 (5) | 4 (4)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 5 (5) | 1 (1) | 11 (11) | 15 (15)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 6 (6) | 4 (4) | 3 (3) | 13 (13) | 5 (5)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 5 (5) | 4 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 6 (6) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 5 (5) | 1 (1) | 9 (9) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 6 (6) | 6 (6) | 6 (6) | 1 (1) | 19 (19) | 9 (9)
Platelet count decreased (Investigations) | 5 (5) | 4 (4) | 4 (4) | 1 (1) | 14 (14) | 6 (6)
Alanine aminotransferase increased (Investigations) | 4 (4) | 5 (5) | 4 (4) | 0 (0) | 13 (13) | 5 (5)
Weight decreased (Investigations) | 3 (3) | 5 (5) | 6 (6) | 0 (0) | 14 (14) | 5 (5)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 4 (4) | 3 (3)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Fatigue (General disorders) | 4 (4) | 5 (5) | 3 (3) | 2 (2) | 14 (14) | 12 (12)
Pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 3 (3)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 7 (7) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Epitaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 4 (4) | 0 (0) | 8 (8) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 2
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 4 (4) | 3 (3) | 2 (2) | 1 (1) | 10 (10) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 5 (5) | 2 (2) | 1 (1) | 10 (10) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
White blood cell count decreased (Investigations) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 6 (6) | 4 (4) | 3 (3) | 13 (13) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 6 (6) | 0
Influenza like illness (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Lip infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 6 (6) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-03): https://cdn.clinicaltrials.gov/large-docs/00/NCT02236000/Prot_SAP_000.pdf